CLINICAL TRIAL: NCT01503281
Title: Effects of Group Vs. Home-Based Combined Exercise-Diet Program In Childhood Obesity: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-UCH-95
Record Dates: First submitted 2012-01-03; First posted 2012-01-04 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: Children; Physical activity; Home-based treatment; Body mass index (z-BMI); Percentage body fat; Waist circumference
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hospital-based exercise program (Experimental): Exercise monitored at the hospital
  Interventions: Other: Circuit training
- Home-based exercise program (Experimental): Participants perform exercise at home
  Interventions: Other: Circuit training
- Control (No Intervention): Control Group participants maintained their usual levels of daily activity, with no additional exercise components.

INTERVENTIONS:
Other: Circuit training — Aerobic and resistance training exercises + Mediterranean diet
  Arms: Home-based exercise program; Hospital-based exercise program

SUMMARY:
The aim of this study was to compare the effect of a hospital group-based vs. home-based combined exercise-diet program for the treatment of childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* overweight/obese

Exclusion Criteria:

* Subjects with severe obesity (z-score above 2.5)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)

PRIMARY OUTCOMES:
Body composition | 6 months
  body mass index (BMI), BMI-Z score

SECONDARY OUTCOMES:
waist circumference | 6 months
Percentage body fat | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU-Cardenal Herrera, Moncada, Valencia, Spain

REFERENCES:
- [Background] Conwell LS, Trost SG, Spence L, Brown WJ, Batch JA. The feasibility of a home-based moderate-intensity physical activity intervention in obese children and adolescents. Br J Sports Med. 2010 Mar;44(4):250-5. doi: 10.1136/bjsm.2008.046359. Epub 2008 May 7. PMID 18463296
- [Background] Watts K, Jones TW, Davis EA, Green D. Exercise training in obese children and adolescents: current concepts. Sports Med. 2005;35(5):375-92. doi: 10.2165/00007256-200535050-00002. PMID 15896088
- [Background] Deforche B, De Bourdeaudhuij I, Debode P, Vinaimont F, Hills AP, Verstraete S, Bouckaert J. Changes in fat mass, fat-free mass and aerobic fitness in severely obese children and adolescents following a residential treatment programme. Eur J Pediatr. 2003 Sep;162(9):616-22. doi: 10.1007/s00431-003-1247-2. Epub 2003 Jun 13. PMID 12811554
- [Derived] Lison JF, Real-Montes JM, Torro I, Arguisuelas MD, Alvarez-Pitti J, Martinez-Gramage J, Aguilar F, Lurbe E. Exercise intervention in childhood obesity: a randomized controlled trial comparing hospital-versus home-based groups. Acad Pediatr. 2012 Jul-Aug;12(4):319-25. doi: 10.1016/j.acap.2012.03.003. Epub 2012 May 26. PMID 22634075
- See also: The University CEU-Cardenal Herrera is the first private University in the Valencian Community. It belongs to the Foundation San Pablo-CEU and is the leading educational organization in Spain with 3 Universities all over Spain. — http://www.uchceu.es